CLINICAL TRIAL: NCT03429829
Title: Fluoride Varnish for Caries Prevention in South African Children: A Cluster-randomized Controlled Community Trial
Brief Title: Fluoride Varnish Community Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DMG Dental Material Gesellschaft mbH (Industry)
Collaborators: Dental Wellness Trust (DWT) (Unknown); University of Western Cape (UWC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Wellflair
Record Dates: First submitted 2018-01-29; First posted 2018-02-12 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Dental Caries; Oral Disease; Costs
Keywords: Caries; Fluoride Varnish; Dental Health; Costs
MeSH Terms: conditions — Dental Caries; Mouth Diseases

STUDY DESIGN:
Intervention Model Description: Children in the reception grade and grade 1 of two schools in a township in South Africa are class-wise cluster-randomized to the fluoride varnish or control groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flairesse varnish (Experimental): Children were part of the LiveSmart tooth brushing program. They all received a new toothbrush at baseline and at every follow-up visit as well as fluoridated toothpaste. Their daily toothbrushing was supervised by the local trained non-professional assistant. In addition, fluoride varnish (22.600 ppm, DMG, Hamburg, Germany) was applied in 3-monthly intervals by the local non-professional assistants who had been trained beforehand and supervised at the first application.
  Interventions: Device: Flairesse varnish
- Control (No Intervention): Children were part of the LiveSmart tooth brushing program. They all received a new toothbrush at baseline and at every follow-up visit as well as toothpaste. Their daily toothbrushing was supervised by the local trained non-professional assistant. Beyond that, the children in this arm were left untreated.

INTERVENTIONS:
Device: Flairesse varnish — Flairesse is applied to enamel and dentine as protective varnish to prevent caries formation and to promote remineralization of initial caries. It is also used in the treatment of hypersensitive teeth by sealing dentin tubules and hypersensitive areas at the neck of the tooth and exposed root dentine. Flairesse varnish contains xylitol and fluoride (22,600 ppm). Both components have been well established for oral health by reducing caries prevalence and incidences.
  During the application, children sat upright; their teeth were first cleaned and dried with cotton wool rolls. After mixing the fluoride varnish, it was applied as a thin layer to all surfaces of the lower and upper dentition, including proximal surfaces (using floss in case of tight contact points) as well as pits and fissures (using a small brush that was provided together with the varnish by the manufacturer). Children were advised not to drink or eat directly after the application, while this could not be controlled.
  Arms: Flairesse varnish

SUMMARY:
This cluster-randomized controlled community trial aimed to assess the efficacy and costs of fluoride varnish application for caries prevention in a high-risk population in South Africa.

DETAILED DESCRIPTION:
Despite advances in oral health, dental caries remains a significant problem - particularly in disadvantaged communities in low- and middle-income countries. A study in the Western Cape Region, which was conducted between 2001 and 2015, reported for example a caries prevalence of 84% for 6-years-old (Smit 2017), highlighting the need for oral health programs and cost-effective interventions. Fluoride varnish offers hereby a feasible possibility to supplement toothbrushing programs in order to improve fluoride delivery and consequently caries prevention. However, many studies failed to confirm the benefits of fluoride varnish for caries prevention, which may partially be explained by the fact that many of these studies were conducted in high-income countries, in which the caries increment is low due to a wide access to fluoride.

This study, thus aimed to further validate the benefits of fluoride varnish application specifically in a primary school setting within a peri-urban, low socio-economic, high-caries risk community in South Africa.

ELIGIBILITY:
Inclusion Criteria:

* Reception grad or grade 1 (age 4-8)
* Signed consent form
* Good general health

Exclusion Criteria:

* Any allergies (especially sticking plaster)
* History of asthma
* Chronic Ulcerated gums
* Chronic Stomatis
* Participation in other study (except LifeSmart)

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 513 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Increment of teeth with cavitated lesions, restorations or extraction. | 2 years
  The primary outcome was the increment of teeth with cavitated lesions (i.e. newly developed ones or progressed, formerly non-cavitated lesions), requiring restorations or extraction.

SECONDARY OUTCOMES:
Increment of teeth with cavitated lesions or restorations. | 2 years
  The increment of teeth with cavitated caries lesions, receiving or requiring a restoration.
Increment of extracted teeth. | 2 years
  The increment of teeth which were extracted due to caries.
Cost | 2 years
  Initial costs of fluoride varnish application and re-treatment costs.

CONTACTS AND LOCATIONS:
Locations (2):
- South Africa (2):
  - Itsitsa Primary School, Mfuleni, Western Cape
  - Nyameko Primary School, Mfuleni, Western Cape

IPD SHARING:
Plan to Share IPD: No